CLINICAL TRIAL: NCT01094847
Title: Clinical Trials to Compare Mosapride Bioavailability Between DWJ1252 and Mosapride Medicine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Somin Bae, Daewoong Pharmaceutical Co. LTD
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_J1252001P
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Bioequivalence

ARMS (3):
- Treatment A (Experimental): DWJ1252 given by oral administration under fasting conditions
  Interventions: Drug: DWJ1252
- Treatment B (Active Comparator): DWJ1252 given by oral administration, 30 minutes after a meal
  Interventions: Drug: DWJ1252
- Treatment C (No Intervention): mosapride by oral administration 30 minutes before meals

INTERVENTIONS:
Drug: DWJ1252 — tablet(oral) administration following the schedule of each arm
  Arms: Treatment A; Treatment B

SUMMARY:
The purpose of this study is to compare and explore bioavailability of mosapride, the main component of DWJ1252(Test drug) and mosapride medicine(Reference drug).

ELIGIBILITY:
Inclusion Criteria:

* a healthy adult male within the range of 20 to 50 years old at the time of screening
* with weight of more than 55kg, in the range of IBW 20%: IBW(kg)={height(cm)-100}*0.9
* who understood completely about this study after the detailed explanation is given, decided to volunteer and gave written informed consent to participate in study in compliance with the requirement of the entire protocol.

Exclusion Criteria:

* one with clinically significant disease in liver, kidney, nerve system, respiratory system, endocrine system, blood, tumor, urinary system, cardiovascular system, mental disease or with medical history
* one with gastrointestinal disease or with gastrointestinal surgical history which can affect the absorption of the investigational drug.
* one with genetic disease like galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
* one who is allergic or has clinically significant allergic history to the component of the investigational drug (mosaprisde), and any component from same family, or to other drugs(Aspirin, antibiotics, etc)
* one who shows different rhythm than sinus rhythm in screening, like QTc >450ms on electrocardiogram, PR interval>200msec or QRS interval 120>msec
* one who shows the following result in clinical laboratory test: AST,ALT>1.25 times of the upper limit of normal range
* one who shows vital signs with the number of systolic blood pressure of 160 mmHg or 100 mmHg, and the number of diastolic blood pressure of 95mmHg or 60mmHg

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Mosapride | 48hr after 1st administration
  AUC(0-last), Cmax

SECONDARY OUTCOMES:
Pharmacokinetics of mosapride, M-1 | 48hr after 1st administration
  * AUCoo, tmax, t 1/2, CL/F, Vd/F of Mosapride
  * AUC(0-last), AUCoo, Cmax, tmax, t 1/2 of M-1

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, Principal Investigator — Seoul National University Hospital IRB
Locations (1):
- Seoul National University Hospital, Seoul, South Korea